CLINICAL TRIAL: NCT02507869
Title: A Pilot Randomized Controlled Trial of an Affect-Guided Physical Activity
Brief Title: A Trial of an Affect-Guided Physical Activity Prescription
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southern Methodist University (Other)
Responsible Party: Principal Investigator, Austin Baldwin, Associate Professor, Southern Methodist University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2012-098-SMIJ
Record Dates: First submitted 2015-07-22; First posted 2015-07-24 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Affect-Guided Prescription (Experimental): Intervention: Participants in the affect-guided condition are instructed to exercise while monitoring how they feel, and to adjust the intensity of their exercise to maintain a pleasant affective response.
  Interventions: Behavioral: Positive affective response
- Heart Rate-Guided Prescription (Active Comparator): Intervention: Participants in the heart rate-guided condition are instructed to exercise while monitoring their heart rate, and to adjust the intensity of the exercise to maintain a heart rate in the moderate range (64-76% of their HRmax).
  Interventions: Behavioral: Moderate-intensity heart rate

INTERVENTIONS:
Behavioral: Positive affective response — Participants adjust the intensity of their exercise to maintain a pleasant affective response.
  Arms: Affect-Guided Prescription
Behavioral: Moderate-intensity heart rate — Participants adjust the intensity of the exercise to maintain a heart rate in the moderate range (64-76% of their HRmax).
  Arms: Heart Rate-Guided Prescription

SUMMARY:
Despite awareness of the benefits of engaging in regular physical activity, at least 50% of adults in the US do not meet recommended guidelines for physical activity. One potential explanation for this lack of regular physical activity is that people often experience exercise as affectively unpleasant. Evidence suggests that the more positively people experience exercise (i.e., the better they feel while exercising), the more likely they are to engage in regular physical activity. This may be especially true for people in poor cardiorespiratory condition. In this randomized trial, investigators compared the effects of an affect-guided exercise prescription (intervention) to a heart rate-guided exercise prescription (control) on change in physical activity minutes among previously underactive adults. Investigators also tested whether the effect of the intervention was moderated by differences in cardiorespiratory fitness.

DETAILED DESCRIPTION:
Regular physical activity has many benefits for overall health and well-being, and current public health guidelines recommend at least 150 minutes per week of moderate-to-vigorous intensity activity to attain these benefits. Despite the many benefits of regular activity, the majority of adults in the US fail to meet recommendations for regular physical activity. One potential explanation for suboptimal levels of physical activity is that exercise is often experienced as affectively unpleasant. Recent work has demonstrated that the more positive people feel during exercise, the more likely they are to engage in regular physical activity. Affective response to exercise is modulated by the intensity of the activity: at a vigorous intensity, affective response is almost uniformly negative and unpleasant, whereas at a moderate intensity, there is more inter-individual variability in affective response. Whether the intensity of the exercise is self-selected or imposed also influences the affective response to exercise, with self-selected intensities being experienced as more pleasant. Current recommendations for engaging in physical activity focus on the type of training intensities most likely to result in a negative affective response. The purpose of this pilot trial was to test the effects of an exercise prescription focused on the maintenance of positive affect during exercise. Investigators randomized participants to one of two exercise prescription conditions: (1) an affect-guided prescription focused on maintaining a positive affective response (intervention), and (2) a heart rate-guided prescription focused on maintaining a moderate intensity (control). Investigators tested the effects of these two exercise prescriptions on changes in subsequent physical activity after one week and one month among a sample of underactive adults. Investigators also tested whether the effect of the intervention was moderated by differences in cardiorespiratory fitness.

ELIGIBILITY:
Inclusion Criteria:

* Physically underactive individuals (< 60 minutes of physical activity/week).

Exclusion Criteria:

* Presence of cardiovascular disease, pulmonary disease, or hypertension.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2013-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change in physical activity minutes measured by the 7-day PAR | One week
Change in physical activity minutes measured by the 7-day PAR | One month

CONTACTS AND LOCATIONS:
Overall Officials: Austin Baldwin, Ph.D., Principal Investigator — Southern Methodist University

REFERENCES:
- [Background] Ekkekakis P, Lind E. Exercise does not feel the same when you are overweight: the impact of self-selected and imposed intensity on affect and exertion. Int J Obes (Lond). 2006 Apr;30(4):652-60. doi: 10.1038/sj.ijo.0803052. PMID 16130028
- [Background] Ekkekakis P, Parfitt G, Petruzzello SJ. The pleasure and displeasure people feel when they exercise at different intensities: decennial update and progress towards a tripartite rationale for exercise intensity prescription. Sports Med. 2011 Aug 1;41(8):641-71. doi: 10.2165/11590680-000000000-00000. PMID 21780850
- [Background] Ekkekakis P, Lind E, Vazou S. Affective responses to increasing levels of exercise intensity in normal-weight, overweight, and obese middle-aged women. Obesity (Silver Spring). 2010 Jan;18(1):79-85. doi: 10.1038/oby.2009.204. Epub 2009 Jun 25. PMID 19556979
- [Background] Parfitt G, Alrumh A, Rowlands AV. Affect-regulated exercise intensity: does training at an intensity that feels 'good' improve physical health? J Sci Med Sport. 2012 Nov;15(6):548-53. doi: 10.1016/j.jsams.2012.01.005. Epub 2012 May 31. PMID 22658587
- [Background] Williams DM, Dunsiger S, Jennings EG, Marcus BH. Does affective valence during and immediately following a 10-min walk predict concurrent and future physical activity? Ann Behav Med. 2012 Aug;44(1):43-51. doi: 10.1007/s12160-012-9362-9. PMID 22532005
- [Background] Williams DM, Dunsiger S, Miranda R Jr, Gwaltney CJ, Emerson JA, Monti PM, Parisi AF. Recommending self-paced exercise among overweight and obese adults: a randomized pilot study. Ann Behav Med. 2015 Apr;49(2):280-5. doi: 10.1007/s12160-014-9642-7. PMID 25223963